CLINICAL TRIAL: NCT00365911
Title: Prevalence of Renal Failure and Risk Factors in an Unreferred Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Prevemed-Medibo (Unknown); Medical Laboratory CRI (Unknown)
Responsible Party: Arjan Van Der Tol, University Hospital Ghent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/038
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: No specific condition
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Taking blood sample — A blood sample will be taken.

SUMMARY:
Blood sample is taken for measurement of serum creatinine, cystatin C, clone V haemoglobin, cholesterol, urine acid, glycemia and CRP.

The medical file is gathered. There will be searched for an association between renal function and cardiovascular risk factors and risk factors by exposition to toxic substantia during work.

ELIGIBILITY:
Inclusion Criteria:

* 20-55 years
* Male and female subjects

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
A possible association between renal clearance and found cardiovascular risk factors and risk factors by exposition to toxic substantia during work. | At time T0

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent; Wim Van Biesen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] van der Tol A, Van Biesen W, Verbeke F, De Groote G, Vermeiren F, Eeckhaut K, Vanholder R. Towards a rational screening strategy for albuminuria: results from the unreferred renal insufficiency trial. PLoS One. 2010 Oct 13;5(10):e13328. doi: 10.1371/journal.pone.0013328. PMID 20967254
- See also: Website University Hospital Ghent — http://www.uzgent.be